CLINICAL TRIAL: NCT01619722
Title: Study of a National Cohort of Adult Patients With Phenylketonuria
Acronym: ECOPHEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRN10/FM-ECOPHEN
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: PKU; Hyperphenylalaninemia
Keywords: PKU; Osteoporosis; HMP; Life quality; Neuropsychological; Nutritial evaluation; Phenylketonuria; Hyperphenylalaninemia
MeSH Terms: conditions — Phenylketonurias; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma an serum at the beginning of study and at 5 years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Phenylketonuria (PKU) is a metabolic disease of genetic origin. This is a rare disease (incidence 1 / 16000 births) which is the subject of a systematic neonatal screening in France, because it is treatable by a diet low in phenylalanine. This plan is required upon confirmation of diagnosis and continued until the age of 8 years. The current trend is to continue the scheme at least until adolescence. Unlike other countries, in France there are no recommendations for a plan "for life". Knowledge about the natural history of PKU in adulthood, the effects of pediatric age, the frequency of complicated shapes, and prognostic factors are poorly documented. On the other hand, there is no consensus on the therapeutic management of this disease in adulthood and monitoring that could be directed towards the detection of neurological disorders and nutrition. Social integration and quality of life of adults PKU patients living in France have not been studied.

DETAILED DESCRIPTION:
The aim off this study is to follow a French cohort of young adult patients with PKU to:

* Describe the evolution of the disease in adulthood and neurological complications associated neuropsychological detect, investigate the prognostic factors for complications
* Describe the metabolic balance of patients
* Collect data on nutritional status,
* Detect osteoporosis
* Studying social integration and quality of life of adult patients with PKU
* Collect biological samples for further study (markers of bone turnover)

Design:

Cohort :

Duration of the inclusion period: 2 years Duration of subject participation: 5 years Total duration of the study: 7 years

JUDGING CRITERIA:

* Complications associated with PKU in adult
* Evolution of neuropsychometric scores
* Bone mineral density by densitometry
* Measuring the quality of life of patients

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Phenylketonuria (PKU) or moderate persistent Hyperphenylalaninemia (HMP) diagnosed by neonatal screening
* Reading and signing an informed consent
* Membership of a social security system

Exclusion Criteria:

* History of severe neurological definite diagnosis could interfere with the detection of neurological disorders associated with PKU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with PKU during a consultation in Hospital care centers.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2012-03-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Evaluate a possible cognitive decline and incidence of neurological complications | 5 years

SECONDARY OUTCOMES:
Determine the prognostic factors of neurological complications | 5 years
  Determine the prognostic factors of these complications, and the impact of the disease and its management on the quality of life (SF-36) and social and professional integration of patients.

CONTACTS AND LOCATIONS:
Overall Officials: François MAILLOT, Pr, Study Director — CHRU TOURS
Locations (16):
- France (16):
  - CHRU-Hôpital Bretonneau - Service de Médecine Interne-Nutrition, Tours, Centre-Val de Loire
  - CHU-ANGERS -Médecine Interne, Angers
  - CHU_Service de Médecine Interne Nutrition A2-Hôpital du Haut Levèque, Bordeaux
  - CHU du Morvan-Département de Pédiatrie et génétique médicale,, Brest
  - Hôpital Femme-Mère-Enfant-Centre de Référence des Maladies Héréditaires du Métabolisme de Lyon, Bron
  - CHU de Dijon--Hôpital des Enfants-Centre de Génétique, Dijon
  - CHU de Grenoble-Hôpital MICHALLON-Unité de Neurologie Générale, Grenoble
  - CHU de LILLE-Hôpital Claude HURIEZ-Service d'Endocrinologie, Lille
  - APHM-Hôpital de la Conception -Médecine Interne, Marseille
  - CHU-Service de Réanimation Pédiatrique / Néonatalogie, Consultation spécialisée en Maladies Héréditaires du Métabolisme, Nantes
  - Hôpital Necker Enfants Malades, APHP-Maladies Métaboliques -Service de Pédiatrie, Paris
  - CHU-RENNES-Hôpital Sud-Service de Génétique-Clinique, Rennes
  - CHU de Rouen-Service de Pédiatrie, Rouen
  - CHU de St Etienne-Hôpital Nord-Service de Pédiatrie, Saint-Etienne
  - CHU-Toulouse-Hôpital PURPAN-Service de Médecine Interne, Toulouse
  - University Hospital of NANCY, Vandœuvre-lès-Nancy